CLINICAL TRIAL: NCT07069088
Title: Clinical Characteristics of Elderly-Onset Versus Adult-Onset Rheumatoid Arthritis; a Cross-Sectional Study
Brief Title: This Study Aims to Characterize and Compare Patients of Adult-onset RA With Patients of Elderly-onset RA Based on the Clinical Manifestations, Disease Activity, Severity Parameters, and Therapeutic Features
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Sara Ahmed Abdelrazik, resident doctor, Sohag University
Other Study IDs: Soh-Med--25-6-5MS
Record Dates: First submitted 2025-06-30; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples to do lab investigations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adult- onset RA group I (16-40 years): 16-40 years
- Adult- onset RA group II (41-60 years): 41-60 years
- EORA >60 years: >60 years

SUMMARY:
This study aims to characterize and compare patients of adult-onset RA with patients of elderly-onset RA based on the clinical manifestations, disease activity, severity parameters, and therapeutic features.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients fulfill the 2010 American College of Rheumatology/ European League Against Rheumatism Classification Criteria for Rheumatoid Arthritis [7] 2) Age of disease onset above 16 years old. 3) patient is cooperative and can answer questions. 4) Patients who are able and willing to give written informed consent.

Exclusion Criteria:

* 1) Other rheumatologic or collagen diseases. 2) Age below 16 years. 3) Active infection 4) Pregnancy 5) Malignancy 6) Uncooperative patients. 7) Patient not able and willing to give written informed consent.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rheumatoid Arthritis patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Disease activity assessment | from enrollment time to the end of examination and investigation at 4 weeks
  Disease activity assessment using DAS 28 Quality of life: HAQ (health assessment questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology and Rehabilitation department at Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patients will be subjected to the following:
  1. Full medical history from the patients, including Demographic data (Age, Sex, Marital status, Occupation, Residence), duration of disease, Comorbidities, and the treatments that patients receive.
  2. Full clinical examination and assessment including:
     1. General examination and Complete rheumatological examination.
     2. Application of American College of Rheumatology/ European League Against Rheumatism Classification Criteria for Rheumatoid Arthritis, on all RA patients.
  3. Laboratory investigations: (Blood sample will be collected into 5ml tubes containing Ethylenediaminetetraacetic acid (EDTA) ).
     * complete blood count (CBC) (done on fully automatic BC 21S hematology analyzer).
     * erythrocyte sedimentation rate (ESR).
     * C- reactive protein (CRP) (using Enzyme-linked immunosorbent assay (ELISA)).
     * rheumatoid factor (RF) (using ELISA).
     * anti-cyclic citrullinated peptide antibody (ACCP Ab) (using ELISA).
  4. Disease activity assessm
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 3 years after the publication of results")
Access Criteria: on clinical trials website

REFERENCES:
- See also: 1. Elderly-onset rheumatoid arthritis — https://pubmed.ncbi.nlm.nih.gov/20554241/